CLINICAL TRIAL: NCT05784363
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Multi-center Exploratory Study to Investigate NT 201 in the Treatment of Enlarged Pores and Excessive Sebum Production in the Face
Brief Title: A Study of NT 201 in the Treatment of Enlarged Pores and Excessive Sebum Production in the Face
Acronym: LESS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M602011077
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Enlarged Pores; Sebum Production
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NT 201 (Experimental): Single NT 201 injection treatment.
  Interventions: Drug: NT 201
- Placebo (Placebo Comparator): Single placebo injection treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NT 201 — Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9 percent (%) Sodium Chloride (NaCl).
  Other Names: IncobotulinumtoxinA; Xeomin/Bocouture®; Xeomin Cosmetic; Xeomeen
  Arms: NT 201
Drug: Placebo — Solution for injection prepared by reconstitution of powder with 0.9% NaCl.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of NT 201 injections in the treatment of enlarged pores and excessive sebum production in the face.

DETAILED DESCRIPTION:
Eligible subjects will be randomized to one of the two treatment groups: NT 201 group and placebo in order to receive one session of injections with either NT 201 or placebo in the upper face (forehead and cheek area) on Day 1 and followed for about 90 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cheek pore size assessed as "large" by the investigator
* Oily skin on the forehead

Exclusion Criteria:

* Treatment with Botulinum toxin (BoNT) of any serotype in the face within the last 12 months
* Facial cosmetic procedure (e.g., chemical peel, photo rejuvenation, mesotherapy, photodynamic therapy, laser treatment, ultrasound treatment, tattooing of eyebrows) within the last 12 months
* Treatment with any dermal filler in the face within the last 12 months
* Any previous insertion of permanent material in the face, including permanent dermal fillers (e.g., silicone, polymethyl methacrylate)
* Any medical condition that may put the subject at increased risk with exposure to botulinum toxin of any serotype

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 4 in Pore Volume in the Cheek Area | Baseline (Day 1), Week 4
  Antera 3D will be used as an assessment tool.
Change from Baseline to Week 4 in Sebum Level in the Forehead Area | Baseline (Day 1), Week 4
  Sebumeter will be used as an assessment tool.

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (3):
- United States (3):
  - Merz Investigation Site #0010473, Los Angeles, California
  - Merz Investigation Site #0010101, Coral Gables, Florida
  - Merz Investigation Site #001097, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No